CLINICAL TRIAL: NCT02509104
Title: An Open-label, Randomized, Single Dose, Two-way Crossover Study to Determine the Bioavailability of One Fixed Dose Combination Capsule Formulation of Dutasteride and Tamsulosin Hydrochloride (0.5 mg/0.2 mg) Relative to Coadministration of One Dutasteride 0.5 mg Capsule and One Tamsulosin Hydrochloride 0.2 mg Tablet in Healthy Male Subjects in the Fed and Fasted States
Brief Title: Bioavailability Study of Fixed Dose Combination (FDC) Dutasteride and Tamsulosin Hydrochloride (HCl) Relative to One Dutasteride and One Tamsulosin HCl Tablet in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 201897
Record Dates: First submitted 2015-07-23; First posted 2015-07-27 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Prostatic Hyperplasia
Keywords: Bioavailability; Dutasteride; Healthy Male Subjects; Fixed Dose Combination
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Dutasteride; Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 Fasted condition (Experimental): Each subject will receive both treatments A and B in either of period 1 or 2 with a washout period of 28 days between treatment periods. Subjects will receive the study treatments under fasting conditions.
  Interventions: Drug: FDC capsule of dutasteride and tamsulosin; Drug: Dutasteride soft gelatine capsule and tamsulosin HCl oral disintegrating tablet
- Cohort 2 Fed condition (Experimental): Each subject will receive both treatment A and B in either of period 1 or 2 with a washout period of 28 days between treatment periods. Subjects will receive the study treatments under fed (high fat breakfast) conditions.
  Interventions: Drug: FDC capsule of dutasteride and tamsulosin; Drug: Dutasteride soft gelatine capsule and tamsulosin HCl oral disintegrating tablet

INTERVENTIONS:
Drug: FDC capsule of dutasteride and tamsulosin — Each FDC capsule contains a mixture of dutasteride formulation (equivalent to 0.5 mg dutasteride) and tamsulosin (equivalent to 0.2 mg tamsulosin) and its physical appearance is hard shell capsule.
Drug: Dutasteride soft gelatine capsule and tamsulosin HCl oral disintegrating tablet — Coadministration of dutasteride soft gelatine capsule and tamsulosin HCl oral disintegrating tablet. Each soft gelatine capsule consist of 0.5 mg of dutasteride and physical appearance is Oblong, size 6, dull yellow capsule. Each oral disintegrating tablet consist of 0.2 mg of tamsulosin and its physical appearance is white, round standard convex.

SUMMARY:
The primary objective of this study is to determine the bioavailability of a FDC capsule formulation of dutasteride and tamsulosin hydrochloride (0.5 milligram [mg]/0.2 mg) relative to coadministration of one dutasteride 0.5 mg capsule and one tamsulosin HCl 0.2 mg tablet in healthy male subjects in fed and fasted states. This is an open-label, randomized, single dose, two-way crossover study enrolling healthy male subjects, split into fasted (Cohort 1) and fed (Cohort 2) conditions. In both cohorts, one FDC capsule formulation of dutasteride 0.5 mg/tamsulosin HCl 0.2 mg will be administered in one treatment period and the coadministration of dutasteride and tamsulosin hydrochloride in a different treatment period. Each subject enrolled will be allowed to participate in only one cohort (i.e, will receive treatment under fasted or fed conditions) and will participate in both treatment periods. The two treatment periods will be separated by a minimum washout period of 28 days. The total duration in the study for each subject will be approximately 2.5 months from screening to the final follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the Medical Monitor if required agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >= 50 kilogram (kg) and body mass index (BMI) within the range 18 to 30 kg per meter square (m^2) (inclusive).
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion Criteria:

* Alanine aminotransferase (ALT) and bilirubin >1.5xUpper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of postural hypotension, dizziness, poor hydration, vertigo, vaso-vagal reactions or any other signs and symptoms of orthostasis, which in the opinion of the investigator could be exacerbated by tamsulosin and result in putting the subject at risk of injury.
* History of diabetes or peptic ulcer disease which is uncontrolled by medical management.
* Current or history of: Breast cancer or clinical breast examination finding suggestive of breast malignancy; Malignancy within the past five years, except for basal cell carcinoma of the skin. Subjects with a prior malignancy who have had no evidence of disease for at least the past 5 years are eligible.
* Prior medical history or evidence of prostate cancer (e.g., positive biopsy, or suspicious ultrasound, or suspicious digital rectal examination [DRE]). Patients with suspicious ultrasound or DRE who have had a negative biopsy within the preceding 6 months and stable prostate specific antigen (PSA) are eligible for the study.
* Based on averaged corrected QT (QTc) values of triplicate ECGs obtained over a brief recording period: QTcF > 450 millisecond (msec).
* Subjects must abstain from taking prescription or non-prescription drugs (including vitamins and dietary or herbal supplements), within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication until completion of the follow-up visit, unless in the opinion of the Investigator and sponsor the medication will not interfere with the Study.
* History of regular alcohol consumption within 6 months of the study defined as: For United States sites: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 gram (g) of alcohol: 12 ounces (360 millilitre [mL]) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL over the duration of the study.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 50 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Unable to swallow and retain oral medication.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-07-30 (Actual); Primary Completion 2015-10-10 (Actual); Study Completion 2015-10-10 (Actual)

PRIMARY OUTCOMES:
Maximum observed serum concentration (Cmax) for dutasteride and tamsulosin | Days 1 to 4 of both treatment periods
  Blood samples for PK analysis will be collected for each subject at the following time points: Pre-dose, 15 minutes (min), 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48 & 72 hours post dose in both the treatment periods. Cmax will be determined for tamsulosin and dutasteride.
Area under the serum concentration-time curve (AUC) zero to time 't' (AUC[0-t]) for tamsulosin and dutasteride; AUC 0 to infinity (AUC 0-inf) will be determined for tamsulosin as data permit | Days 1 to 4 of both treatment periods
  Blood samples for PK analysis will be collected for each subject at the following time points: Pre-dose, 15 minutes (min), 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48 & 72 hours post dose in both the treatment periods. AUC 0-t will be determined for tamsulosin and dutasteride. Additionally, AUC 0-inf will be determined for tamsulosin as data permit.

SECONDARY OUTCOMES:
Time of occurrence of Cmax (Tmax) for dutasteride and tamsulosin | Days 1 to 4 of both treatment periods
  Blood samples for PK analysis will be collected for each subject at the following time points: Pre-dose, 15 minutes (min), 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48 & 72 hours post dose in both the treatment periods. Tmax will be determined for tamsulosin and dutasteride.
Terminal phase half-life (t1/2) for tamsulosin | Days 1 to 4 of both treatment periods
  Blood samples for PK analysis of tamsulosin and dutasteride will be collected for each subject at the following time points: Pre-dose, 15 minutes (min), 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48 & 72 h post dose in both the treatment periods. Terminal phase half-life will be determined for tamsulosin.
Number of participants with adverse events (AE) /serious adverse event (SAE) as a measure of safety and tolerability | From start of study treatment until follow-up contact (up to Week 7)
  AEs and SAEs will be collected from the start of study Treatment until the follow-up contact.
Composite of vital signs as a measure of safety and tolerability | Screening visit, Day -1, and Day 2 (in both treatment periods) and follow-up visit (up to 2.5 months).
  Vital signs will be measured in semi-supine position after 5 minutes rest and will include temperature, systolic and diastolic blood pressure and pulse rate.
Composite of 12-lead electrocardiogram (ECG) assessment as a safety measure | Screening, Day 1 and Day 2 in both treatment periods and follow-up visit (up to 2.5 months).
  ECG measurement include heart rate and measures PR, QRS, QT, and QT interval corrected using the Fridericia's formula (QTcF) intervals.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Burns O, Zhu J, Manyak MJ, Ravindranath R, Koosha F, Haque N, Chung S. Relative Bioavailability of Fixed-Dose Combinations of Tamsulosin and Dutasteride: Results From 2 Randomized Trials in Healthy Male Volunteers. Clin Pharmacol Drug Dev. 2018 May;7(4):422-434. doi: 10.1002/cpdd.380. Epub 2017 Aug 11. PMID 28800206
- See also: Results for study 201897 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/201897?search=study&search_terms=201897#rs
- Available data/document: Clinical Study Report: 201897 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 201897 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 201897 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 201897 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 201897 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 201897 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 201897 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register